CLINICAL TRIAL: NCT03296124
Title: Prognostic Value of Androgen Receptor Expression and Mutations Within Oncogenes and Tumor Suppressor Genes in Patients Treated for High Risk Prostate Cancer With Proton Therapy
Brief Title: Prognostic Value of Androgen Receptor Expression and Mutations Within Oncogenes and Tumor Suppressor Genes in Patients Treated for High Risk Prostate Cancer With Proton Therapy (PRX32)
Acronym: PRX32
Status: Withdrawn | Type: Observational
Why Stopped: This project currently does not have any subjects enrolled due to other PI priorities.
Sponsor: University of Florida (Other)
Collaborators: Driver (Unknown)
Responsible Party: Sponsor
Other Study IDs: UFPTI 1612- PRX32; IRB201700018 (Other: UF IRB)
Record Dates: First submitted 2017-09-14; First posted 2017-09-28 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Proton Radiation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective Review Study for Prognostic Transcriptional Output Related to Androgen Receptor Expression in Patients Treated for High Risk Prostate Cancer with Proton Therapy

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (older than 18 years at time of treatment) with high risk prostate cancer who were treated with proton therapy at UFHPTI/Department of Radiation Oncology
* Patients treated between 6/10/2010 through 4/26/17 with at least 2 years follow up

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion (target study population) criteria for this retrospective outcomes analysis are adult patients (older than 18 years at time of treatment) with high risk prostate cancer who were treated with proton therapy at UFHPTI/Department of Radiation Oncology. For this retrospective outcomes study, data will be used from patients treated between 6/10/2010 through 4/26/17 with at least 2 years follow up.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemistry of tumor cell proteins will be performed on prostate biopsies to detect for androgen receptors and other protein products related to oncogenes or tumor suppressor genes thought to play a role in radiation or ADT. | 2 years follow up

SECONDARY OUTCOMES:
DNA sequencing will be performed on prostate tumor DNA to determine the mutational status of several oncogenes and tumor suppressor genes including genes coding androgen receptors. | 2 years follow up
RNA sequencing will be performed on several oncogenes and tumor suppressor genes including genes coding androgen receptors to detect RNA expression including genes related to the androgen receptor. | 2 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Curtis M Bryant, MD, MPH, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The collection of sensitive information about subjects is limited to the amount necessary to achieve the aims of the research, so that no unneeded sensitive information is being collected.

REFERENCES:
- [Background] Roach M 3rd, Bae K, Speight J, Wolkov HB, Rubin P, Lee RJ, Lawton C, Valicenti R, Grignon D, Pilepich MV. Short-term neoadjuvant androgen deprivation therapy and external-beam radiotherapy for locally advanced prostate cancer: long-term results of RTOG 8610. J Clin Oncol. 2008 Feb 1;26(4):585-91. doi: 10.1200/JCO.2007.13.9881. Epub 2008 Jan 2. PMID 18172188
- [Background] Denham JW, Steigler A, Lamb DS, Joseph D, Turner S, Matthews J, Atkinson C, North J, Christie D, Spry NA, Tai KH, Wynne C, D'Este C. Short-term neoadjuvant androgen deprivation and radiotherapy for locally advanced prostate cancer: 10-year data from the TROG 96.01 randomised trial. Lancet Oncol. 2011 May;12(5):451-9. doi: 10.1016/S1470-2045(11)70063-8. PMID 21440505
- [Background] Sydes MR, Stephens RJ, Moore AR, Aird EG, Bidmead AM, Fallowfield LJ, Graham J, Griffiths S, Mayles WP, McGuire A, Stanley S, Warrington AP, Dearnaley DP; RT01 collaborators. Implementing the UK Medical Research Council (MRC) RT01 trial (ISRCTN 47772397): methods and practicalities of a randomised controlled trial of conformal radiotherapy in men with localised prostate cancer. Radiother Oncol. 2004 Aug;72(2):199-211. doi: 10.1016/j.radonc.2004.04.007. PMID 15297138
- [Background] Liauw SL, Weichselbaum RR, Rash C, Correa D, Al-Hallaq HA, Pelizzari CA, Jani AB. Biochemical control and toxicity after intensity-modulated radiation therapy for prostate cancer. Technol Cancer Res Treat. 2009 Jun;8(3):201-6. doi: 10.1177/153303460900800304. PMID 19445537
- [Background] D'Amico AV, Chen MH, Renshaw AA, Loffredo M, Kantoff PW. Androgen suppression and radiation vs radiation alone for prostate cancer: a randomized trial. JAMA. 2008 Jan 23;299(3):289-95. doi: 10.1001/jama.299.3.289. PMID 18212313
- [Background] Christensen M, Najy AJ, Snyder M, Movilla LS, Kim HR. A critical role of the PTEN/PDGF signaling network for the regulation of radiosensitivity in adenocarcinoma of the prostate. Int J Radiat Oncol Biol Phys. 2014 Jan 1;88(1):151-8. doi: 10.1016/j.ijrobp.2013.10.019. PMID 24331662
- [Background] Paximadis P, Najy AJ, Snyder M, Kim HR. The interaction between androgen receptor and PDGF-D in the radiation response of prostate carcinoma. Prostate. 2016 May;76(6):534-42. doi: 10.1002/pros.23135. Epub 2016 Jan 6. PMID 26732854
- [Background] Mettlin CJ, Murphy GP, Rosenthal DS, Menck HR. The National Cancer Data Base report on prostate carcinoma after the peak in incidence rates in the U.S. The American College of Surgeons Commission on Cancer and the American Cancer Society. Cancer. 1998 Oct 15;83(8):1679-84. doi: 10.1002/(sici)1097-0142(19981015)83:83.0.co;2-y. PMID 9781963
- [Background] Spratt DE, Pei X, Yamada J, Kollmeier MA, Cox B, Zelefsky MJ. Long-term survival and toxicity in patients treated with high-dose intensity modulated radiation therapy for localized prostate cancer. Int J Radiat Oncol Biol Phys. 2013 Mar 1;85(3):686-92. doi: 10.1016/j.ijrobp.2012.05.023. Epub 2012 Jul 12. PMID 22795805
- [Background] Vora SA, Wong WW, Schild SE, Ezzell GA, Andrews PE, Ferrigni RG, Swanson SK. Outcome and toxicity for patients treated with intensity modulated radiation therapy for localized prostate cancer. J Urol. 2013 Aug;190(2):521-6. doi: 10.1016/j.juro.2013.02.012. Epub 2013 Feb 13. PMID 23415964
- [Background] Horwitz EM, Bae K, Hanks GE, Porter A, Grignon DJ, Brereton HD, Venkatesan V, Lawton CA, Rosenthal SA, Sandler HM, Shipley WU. Ten-year follow-up of radiation therapy oncology group protocol 92-02: a phase III trial of the duration of elective androgen deprivation in locally advanced prostate cancer. J Clin Oncol. 2008 May 20;26(15):2497-504. doi: 10.1200/JCO.2007.14.9021. Epub 2008 Apr 14. PMID 18413638
- [Background] Bartek J, Mistrik M, Bartkova J. Androgen receptor signaling fuels DNA repair and radioresistance in prostate cancer. Cancer Discov. 2013 Nov;3(11):1222-4. doi: 10.1158/2159-8290.CD-13-0679. PMID 24203954
- [Background] Polkinghorn WR, Parker JS, Lee MX, Kass EM, Spratt DE, Iaquinta PJ, Arora VK, Yen WF, Cai L, Zheng D, Carver BS, Chen Y, Watson PA, Shah NP, Fujisawa S, Goglia AG, Gopalan A, Hieronymus H, Wongvipat J, Scardino PT, Zelefsky MJ, Jasin M, Chaudhuri J, Powell SN, Sawyers CL. Androgen receptor signaling regulates DNA repair in prostate cancers. Cancer Discov. 2013 Nov;3(11):1245-53. doi: 10.1158/2159-8290.CD-13-0172. Epub 2013 Sep 11. PMID 24027196
- [Background] Raghu D, Paul PJ, Gulati T, Deb S, Khoo C, Russo A, Gallo E, Blandino G, Chan AL, Takano E, Sandhu SK, Fox SB, Williams S, Haupt S, Gamell C, Haupt Y. E6AP promotes prostate cancer by reducing p27 expression. Oncotarget. 2017 Jun 27;8(26):42939-42948. doi: 10.18632/oncotarget.17224. PMID 28477016
- [Background] Malla B, Zaugg K, Vassella E, Aebersold DM, Dal Pra A. Exosomes and Exosomal MicroRNAs in Prostate Cancer Radiation Therapy. Int J Radiat Oncol Biol Phys. 2017 Aug 1;98(5):982-995. doi: 10.1016/j.ijrobp.2017.03.031. Epub 2017 Mar 27. PMID 28721912
- [Background] Bostrom PJ, Bjartell AS, Catto JW, Eggener SE, Lilja H, Loeb S, Schalken J, Schlomm T, Cooperberg MR. Genomic Predictors of Outcome in Prostate Cancer. Eur Urol. 2015 Dec;68(6):1033-44. doi: 10.1016/j.eururo.2015.04.008. Epub 2015 Apr 23. PMID 25913390
- [Background] Choudhury AD, Eeles R, Freedland SJ, Isaacs WB, Pomerantz MM, Schalken JA, Tammela TL, Visakorpi T. The role of genetic markers in the management of prostate cancer. Eur Urol. 2012 Oct;62(4):577-87. doi: 10.1016/j.eururo.2012.05.054. Epub 2012 Jun 5. PMID 22695242
- See also: Cancer Facts & Figures 2017. 2017. Atlanta, GA: American Cancer Society. — https://www.cancer.org/research/cancer-facts-statistics/all-cancer-facts-figures/cancer-facts-figures-2017.html